CLINICAL TRIAL: NCT07197372
Title: Efficacy of Sacubitril/Valsartan Versus Captopril in Children With Dilated Cardiomyopathy Admitted to Assiut University Children Hospital: A Prospective Comparative Cohort Study
Brief Title: Comparative Efficacy of ARNI Versus ACE Inhibitor Therapy in Egyptian Children With Dilated Cardiomyopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Jehan Hani Zein El-Abidin Hussein, resident doctor at pediatrics department, Assiut University
Other Study IDs: Valsartan vs. Captopril
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: ARNI; Pediatric Dilated Cardiomyopathy; ACE Inhibitor
Keywords: ARNI; pediatric dilated cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The population consists of Egyptian pediatric patients aged 1 month to 18 years who have been diagno: Eligible patients must demonstrate echocardiographic evidence of ventricular dilation (LVEDD z-score >2) and systolic dysfunction (LVEF <45%, FS <25%). They are required to be clinically stable, on conventional background therapy, but not previously treated with sacubitril/valsartan or captopril. Children with other cardiomyopathy forms, severe renal or hepatic impairment, or significant electrolyte imbalance are excluded. The study will include a balanced distribution of both sexes, across pediatric age groups (ranging from infants to adolescents), reflective of the typical spectrum of DCM presentation in Egypt.

SUMMARY:
This is a prospective, cohort study designed to evaluate the efficacy and safety of sacubitril/valsartan versus captopril in children with dilated cardiomyopathy (DCM) admitted to Assiut University Children Hospital over a one-year period.

DETAILED DESCRIPTION:
The trial aims to directly compare two therapies for pediatric dilated cardiomyopathy. Captopril, an ACE inhibitor, has long been the gold standard in managing pediatric heart failure. However, sacubitril/valsartan, an angiotensin receptor-neprilysin inhibitor (ARNI), has emerged as a potentially superior therapy with demonstrated benefits in adults. This study will assess if the newer ARNI therapy provides improved cardiac function and tolerability compared to traditional ACE inhibition in Egyptian children with DCM. Children meeting echocardiographic diagnostic criteria for systolic dysfunction will be randomized into two treatment arms. Over twelve months, detailed clinical, echocardiographic, and laboratory evaluations will track changes in left ventricular ejection fraction (LVEF), hospitalizations, safety, and quality of life. The ultimate goal is to establish evidence-based guidance for the optimal treatment of pediatric DCM in Egypt.electrolyte imbalance are excluded. The study will include a balanced distribution of both sexes, across pediatric age groups (ranging from infants to adolescents), reflective of the typical spectrum of DCM presentation in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 month to 18 years

Diagnosed with dilated cardiomyopathy via echocardiography

LVEDD z-score > 2 (indexed to body surface area or age)

LVEF <45% and FS <25%

Clinically stable for ≥2 weeks prior to enrollment

Receiving optimized guideline-based heart failure therapy (excluding ACEI/ARNI prior to study)

Exclusion Criteria:

* Known hypersensitivity/contraindications to ACEIs or ARNIs

Severe renal impairment (eGFR <30 mL/min/1.73 m²)

Persistent hyperkalemia (K+ >5.5 mmol/L)

Other cardiomyopathies (hypertrophic, restrictive) or unrelated congenital/structural heart disease

Severe hepatic impairment

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible patients must demonstrate echocardiographic evidence of ventricular dilation (LVEDD z-score >2) and systolic dysfunction (LVEF <45%, FS <25%). They are required to be clinically stable, on conventional background therapy, but not previously treated with sacubitril/valsartan or captopril. Children with other cardiomyopathy forms, severe renal or hepatic impairment, or significant electrolyte imbalance are excluded. The study will include a balanced distribution of both sexes, across pediatric age groups (ranging from infants to adolescents), reflective of the typical spectrum of DCM presentation in Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-05-30 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fractio | one year
  LVEF is measured using pediatric echocardiography at baseline and after 12 months. Improvement or decline in LVEF will be used to directly compare therapeutic efficacy.

IPD SHARING:
Plan to Share IPD: No